CLINICAL TRIAL: NCT04349202
Title: Beaumont Health Large-scale Automated Serologic Testing for COVID-19
Acronym: BLAST COVID-19
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Matthew Sims, MD, PhD, Director Infectious Disease Research, Beaumont Health; Professor of Internal Medicine and Foundational Medical Studies, OUWB School of Medicine, Corewell Health East
Other Study IDs: 2020-134
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: COVID-19; Coronavirus Infection; Severe Acute Respiratory Syndrome Coronavirus 2
Keywords: Exposure, Occupational; COVID-19 virus infection; COVID-19 pandemic; COVID-19 virus testing; SARS-CoV-2 antibodies
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Beaumont employees: Beaumont employees (employees and affiliated non-employed physicians and advanced practice providers) undergoing serology testing for SARS-CoV-2 antibodies, their immediate family members, and members of other high-risk groups.
  Interventions: Diagnostic Test: EUROIMMUN assay

INTERVENTIONS:
Diagnostic Test: EUROIMMUN assay — Serology testing to detect SARS-CoV-2 antibodies

SUMMARY:
The purpose of this study is to determine how peoples' bodies respond to exposure to COVID-19. Employees of Beaumont Health in Michigan who are older than 18 years may be eligible to participate. Participants from other high-risk groups who are not Beaumont employees may also be recruited, as may family members of Beaumont employees who have tested positive for COVID-19. Participants will have blood drawn two or more times for serology testing. This serology test will determine if participants have detectable levels of the antibodies that our bodies develop to fight COVID-19 infection. Participants will fill out a questionnaire each time they provide a blood sample. The questionnaires include questions about participants' personal traits; their health; general questions about their risk to exposure; job and risk of exposure; symptoms, diagnosis, treatment of COVID-19 since last blood draw. Researchers will monitor participants' medical records in a confidential manner for one year after the last blood draw to help determine if people who develop antibodies to COVID-19 are protected against developing a COVID-19 infection in the future.There may be no direct benefits for participants; however, information from this study may benefit other people by increasing our understanding of COVID-19, how it spreads from person to person, and how people respond to fight off the infection.The results of the serology test are used for research only and will not affect clinical decisions regarding participants' treatment or quarantine

DETAILED DESCRIPTION:
Beaumont Health is an eight-hospital regional health care system with a total of 3,337 beds, 38,000 employees and 5,000 physicians in Southeast Michigan. In the first 3 weeks of the COVID-19 pandemic within Michigan over 3300 patients tested positive through our system and over 1000 have been admitted for inpatient care. COVID-19 has a wide range of presentations from asymptomatic to multisystem organ failure and death. Spread from asymptomatic individuals has been described in the literature but the extent of this transmission is unclear. Large scale serologic testing can help address this question by detecting antibodies generated after an individual is infected with COVID-19. Healthcare workers have developed COVID-19 but the true infection rate among those who care for COVID-19 patients and whether the infection occurs at work is unknown.

Every day, thousands of Beaumont physicians, nurses, technicians and other caregivers are working under extraordinary stress, doing their very best to care for patients with this highly contagious and potentially deadly virus. They are trying to protect themselves from infection while dealing with personal protective equipment requirements and limited knowledge of who in the hospital environment may be carrying the infection and potentially spreading it among the staff. Caregivers are at greater risk of infection than the public, and when they become sick, it reduces the number of trained personnel available to care for hospitalized patients. Serological testing would give Beaumont's front-line staff, family members and patients peace of mind by determining infection rates in our care units. Knowing the infection rates will demonstrate how effective the use of personal protective equipment has been for staff, whether any flaws exist in the system, and how many clinical staff currently have potentially protective antibodies.

Beaumont Health has 2 EURO Lab Workstations capable of running the SARS-CoV-2 IgG and IgA EUROIMMUN serology assay (referred to as the EUROIMMUN assay hereafter). Each EUROIMMUN assay consists of 2 separate tests; one of which measures IgG (the memory antibody which should give long acting resistance to people who mount an immune response) and the second of which measures IgA (the secretory antibody that should protect against infection through mucous membranes). Researchers can run 5,000 samples a day with each sample being tested for IgA and IgG.

Potential participants (employees and affiliated non-employed physicians and advanced practice providers) will provide informed consent. Researchers will analyze all participants over 2 blood draws between 2 and 4 weeks apart to see if they developed antibodies to COVID-19. Participants at medium risk for exposure in their job function at Beaumont will have 3 draws 2-4 weeks apart and people considered the highest risk, those who provide the direct patient care to COVID-19 patients, will be tested 2-4 weeks apart until the pandemic in Michigan is under control (estimated to be 8 blood draws). If the participants agree, researchers will bank 0.5 ml of serum for future testing related to COVID-19. An initial questionnaire and subsequent questionnaires with each blood draw will be completed by participants. Biostatistics will analyze the data from the questionnaires and the serology test to determine any links between level of risk associated with the participants job, medical history, and exposure history to development of COVID-19 antibodies. Participants medical records will be monitored for one year to see if they are diagnosed with COVID-19 and if they have a positive PCR test for COVID-19 since they were tested for the presence of antibodies. All employees identified as developing COVID-19 after their antibody levels were tested will be analyzed and a correlation between antibody level and development of COVID-19 will be generated. This will allow an estimation of the protective effect of antibodies relative to people who have no detectable antibodies. Researchers will perform an epidemiologic analysis to identify contacts between staff and patients based on records in the EMR and can cross reference to determine if nosocomial transmission is likely occurring from staff to patients and vice versa. Researchers will also determine if there was any likely exposure to patients with COVID-19 on the same floor or if prior patients in the room had COVID-19. This will also allow researchers to model the rate of spread of the virus within the hospital from unknown sources.

Additional studies on subpopulations of participants will test whether antibody tests on dried blood spots (small drops of blood applied to filter paper, which do not have to be refrigerated) correlate with results obtained from drawing a full vial of blood. Reproducibility, stability, the effect of shipping, inter-lab concordance and any differences between participant-collected and phlebotomist-collected blood spot samples will be tested.

An additional subpopulation study will test immediate family members of participants who test positive for SARS-CoV-2 antibodies to evaluate intra-family spread of the disease. Another subpopulation study will recruit participants from other high-risk populations at the discretion of the investigators.

ELIGIBILITY:
Inclusion Criteria:

* Beaumont Health employees and affiliated non-employed physicians and advanced practice providers
* Immediate family members of Beaumont Health employees, affiliated non-employed physicians and advance practice providers who have tested positive for SARS-CoV-2 antibodies
* non-Beaumont employees who are specifically invited to participate in the study by Dr. Sims, Dr. Kennedy, or Dr. Maine
* All ages

Exclusion Criteria:

* Decisionally impaired
* Individuals symptomatic for COVID-19 <72 hours prior to testing appointment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Beaumont Health Employees and affiliated non-employed physicians and advanced practice providers
  Immediate family members of Beaumont Health employees, affiliated non-employed physicians and advance practice providers who have tested positive for SARS-CoV-2 antibodies
  Members of other high-risk populations as determined by the investigators who are specifically invited by Dr. Sims, Dr. Kennedy or Dr. Maine
Sampling Method: Non-Probability Sample
Enrollment: 20614 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

PRIMARY OUTCOMES:
Prevalence COVID antibodies in employees of Beaumont Health | 1 year
  Number of participants testing positive for the presence of IgG or IgA antibodies to SARS-CoV-2 using the EUROIMMUN Serology testing platform. Serology testing of Beaumont Health employees will allow an estimation of asymptomatic carriage and help determine level of nosocomial spread of COVID-19 within our institution among its employees. All participants will provide a minimum of 2 blood draws between 2 and 4 weeks apart to determine the presence of antibodies to COVID-19. Participants at medium risk for exposure in their job function at Beaumont will have 3 draws 2-4 weeks apart and people considered the highest risk, those who provide the direct patient care to COVID-19 patients, will be tested 2-4 weeks apart until the pandemic in Michigan is under control (estimated to be 8 blood draws).

SECONDARY OUTCOMES:
COVID-19 re-infection in participants positive for antibodies to SARS-CoV-2 | 1 year
  Number of participants with positive detection of anti-SARS-CoV-2 antibodies using the EUROIMMUN Serology testing platform, who later develop a COVID-19 infection as documented in Beaumont Health electronic medical records
Correlation of dried blood spot and standard blood sampling positive for COVID-19 IgG antibodies | 1 yr
  Number of participants with positive SARS-CoV-2 serum IgG antibodies using the EUROIMMUN Serology testing platform from standard collection of 1 vial (approximately 5ml) of blood who also test positive for anti-SARS-CoV-2 IgG antibodies using dried blood spot samples
Correlation of dried blood spot and standard blood sampling negative for COVID-19 IgG antibodies | 1 yr
  Number of participants with negative SARS-CoV-2 serum IgG antibodies using the EUROIMMUN Serology testing platform from standard collection of 1 vial (approximately 5ml) of blood who also test negative for anti-SARS-CoV-2 IgG antibodies using dried blood spot samples
Correlation of dried blood spot and standard blood sampling positive for COVID-19 IgA antibodies | 1 yr
  Number of participants with positive SARS-CoV-2 serum IgA antibodies using the EUROIMMUN Serology testing platform from standard collection of 1 vial (approximately 5ml) of blood who also test positive for anti-SARS-CoV-2 IgA antibodies using dried blood spot samples
Correlation of dried blood spot and standard blood sampling negative for COVID-19 IgA antibodies | 1 yr
  Number of participants with negative SARS-CoV-2 serum IgA antibodies using the EUROIMMUN Serology testing platform from standard collection of 1 vial (approximately 5ml) of blood who also test negative for anti-SARS-CoV-2 IgA antibodies using dried blood spot samples
Reproducibility of SARS-CoV-2 IgG antibody detection from dried blood spots | 1 yr
  Number of participants with identical SARS-CoV-2 IgG antibody results using the EUROIMMUN Serology testing platform from separate blood spot samples collected on the same day
Stability of dried blood spots for SARS-CoV-2 IgG antibody detection | 1 year
  Number of participants with identical SARS-CoV-2 IgG antibody results using the EUROIMMUN Serology testing platform from blood spots collected on the same day but tested after 7 to 28 days of storage
Effect of shipping on dried blood spot samples for SARS-CoV-2 IgG antibody detection | 1 yr
  Number of participants with identical SARS-CoV-2 IgG antibody results using the EUROIMMUN Serology testing platform from dried blood spot samples processed at Beaumont Health and those shipped to EUROIMMUN (Lubeck, Germany) for testing
Accuracy of participant-performed blood spot collection for SARS-CoV-2 IgG antibody detection | 1 yr
  Number of participants with identical SARS-CoV-2 IgG antibody results using the EUROIMMUN Serology testing platform from dried blood spot samples collected by a phlebotomist and those self-collected by the participant using an instructional information sheet
Ease of participant-performed blood spot collection | 1 yr
  Ease of following an instructional information sheet to self-collect blood spots will be rated by the participant on a 10 point scale where 1 indicates complete comfort and understanding the collection procedure and 10= extreme difficulty with understand the information sheet and collecting blood spots
Correlation of SARS-CoV-2 antibodies between immediate family members | 1 yr
  Number of immediate family member participants testing positive for SARS-CoV-2 IgG antibodies using the EUROIMMUN Serology testing platform following a SARS-CoV-2 IgG antibody positive assay in a Beaumont Health employee participant

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Sims, MD, PhD, Principal Investigator — Corewell Health East
Locations (2):
- United States (2):
  - Beaumont Health System, Royal Oak, Michigan
  - Beaumont Health, Royal Oak, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sims MD, Podolsky RH, Childers KL, Higgins B, Trueman J, Homayouni R, Voss DR, Berkiw-Scenna N, Keil H, Kennedy RH, Maine GN. Dried blood spots are a valid alternative to venipuncture for COVID-19 antibody testing. J Immunol Methods. 2023 Feb;513:113420. doi: 10.1016/j.jim.2022.113420. Epub 2022 Dec 31. PMID 36596443
- [Derived] Sims MD, Maine GN, Childers KL, Podolsky RH, Voss DR, Berkiw-Scenna N, Oh J, Heinrich KE, Keil H, Kennedy RH, Homayouni R. Coronavirus Disease 2019 (COVID-19) Seropositivity and Asymptomatic Rates in Healthcare Workers Are Associated with Job Function and Masking. Clin Infect Dis. 2021 Jul 30;73(Suppl 2):S154-S162. doi: 10.1093/cid/ciaa1684. PMID 33150375